CLINICAL TRIAL: NCT06877013
Title: An Exploratory, Randomized, Single Blinded, Monocentric, Parallel Group Study to Explore the Tolerance Profile of Soluble Fibers in Individuals With Self-perceived Gastrointestinal Sensitivity to Fibers
Brief Title: Tolerance Profile of Soluble Fibers in Individuals With Self-perceived GI Sensitivity to Fibers (Tarine)
Acronym: Tarine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 23REX0061999
Record Dates: First submitted 2025-02-17; First posted 2025-03-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Population With Self-perceived Gastro-intestinal Sensitivity to Fibers
Keywords: Exploratory; Monocentric; Single blinded; Randomized; Multi-dose; Soluble fibers; Gastro-intestinal sensitivity; Parallel study; Placebo-challenge

STUDY DESIGN:
Intervention Model Description: Single blinded, Randomized, Parallel group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose 1 (Experimental): 8.0g oligosaccharide FODMAP A + 1.6g oligosaccharide FODMAP B
  Interventions: Other: Fiber's mix (among 4 doses)
- Dose 2 (Experimental): 12g oligosaccharide FODMAP A + 2.4g oligosaccharide FODMAP B
  Interventions: Other: Fiber's mix (among 4 doses)
- Dose 3 (Experimental): 16g oligosaccharide FODMAP A + 3.2g oligosaccharide FODMAP B
  Interventions: Other: Fiber's mix (among 4 doses)
- Dose 4 (Experimental): 20g oligosaccharide FODMAP A + 4.0g oligosaccharide FODMAP B
  Interventions: Other: Fiber's mix (among 4 doses)
- Placebo (Experimental): 8.0 g Dextrose
  Interventions: Other: Placebo challenge

INTERVENTIONS:
Other: Placebo challenge — 2 sachets per day over 7-day challenge
  Arms: Placebo
Other: Fiber's mix (among 4 doses) — 2 sachets per day over 7-day challenge
  Arms: Dose 1; Dose 2; Dose 3; Dose 4

SUMMARY:
The purpose of this study is to determine the optimal dose of soluble fibers that induces tolerable gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years of age inclusive, and Body Mass Index (BMI) 18.5-29.9 kg/m2 inclusive; who according to the Rome IV fulfil criteria for self-perceived sensitivity to fructans and/or α-GOS including subjects diagnosed with IBS, FBFB, or FBD-U.
2. 18-60 years of age inclusive, and BMI 18.5-29.9 kg/m2 inclusive; who fulfil criteria for self-perceived sensitivity to oligosaccharide FODMAP A and B, not diagnosed with IBS, FB or FBD-U as per Rome IV Criteria but reporting abdominal pain once a week AND/OR bloating/distention once a week as per ROME IV diagnostic questionnaire.
3. Individuals who fully understand the objectives of the study, who are willing to provide consent and agree to follow the protocol of the study.
4. Subject is covered by French health insurance.
5. Subject agrees to be registered in the national database of subjects participating in clinical research.
6. Subject is willing and able to complete the electronic Patient Reported Outcomes (ePRO) using their digital device (e.g. smartphone) having access to internet (web site).
7. Female subjects must either be postmenopausal for at least 12 months or have undergone specific surgical procedures resulting in sterility (such as hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or they are using one of the medically approved contraceptive methods listed below from V1 until the end of the study, such as, but not exclusively:

   * Oral contraception
   * Intra-uterine device (IUD)
   * Double barrier method (e.g., condoms and spermicide)
   * Abstinence, when the opinion of the investigator, their occupation or lifestyle gives efficient evidence that abstinence will be maintained throughout the study and for one month thereafter.

Exclusion Criteria:

1. Individuals who score above 300 on the Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) if diagnosed with IBS using the Rome IV criteria.
2. Individuals that are diagnosed with any other chronic gastrointestinal disease or condition including inflammatory bowel disease, coeliac disease, fistulas or physiological/mechanical gastrointestinal obstruction, diverticulitis, gastric bezoar, radiation enteritis, suspected or known strictures.
3. Change of dietary habits within the 4 weeks preceding V1 (e.g., start of a diet rich in fibers) or planned change (e.g., start of a new diet during study participation).
4. Individuals with specific and extreme diets (e.g.: strict low-FODMAP, gluten free, high fiber diet, etc.).
5. Individuals who anticipate changes to consumption of naturally probiotic/prebiotic containing foods e.g., yogurt with live cultures etc., in the next 2 months.
6. Subject who has planned to participate in another clinical study during the period of this study OR subject involved in any other clinical study in the past four weeks.
7. Subject with known allergy to any component of the study product(s).
8. Individuals receiving any form of treatment likely to interfere with metabolism or dietary habits (e.g., anorexia, weight loss.).
9. Subject with any intake of antibiotics or intestinal antiseptics in the previous month (within 30 days) prior to screening visit (V1).
10. Individuals with current use of medication with central nervous system effects as judged by the investigator.
11. Individuals with previous digestive surgery (except for appendectomy and cholecystectomy performed more than 2 years ago).
12. Subjects performing strenuous daily exercise for more than 1.5 hours at a time (e.g., intensive daily cardio for more than 1.5 hours).
13. Oral disease that may impact on hydrogen and methane breath sampling e.g., gingivitis, halitosis, oral thrush, candidiasis.
14. Subject with any intake of drugs that might modify gastrointestinal function (e.g., regular use of laxatives, anti-diarrheal agents, anti-emetics, prokinetics, proton pump inhibitors (PPIs), NSAIDs, antacids, etc.).
15. Individuals who take supplements used to treat bloating: activated charcoal, enzymes (ex: lactase, alpha galactosidase, fructanase).
16. Women who report they are pregnant/lactating/planning pregnancy.
17. Recent/ongoing consumption of probiotics/prebiotic supplements (past 28 days).
18. Subject is a smoker (use of any tobacco products, nicotine, or nicotine-containing products in the previous 3 months).
19. Alcohol consumption that exceeds the recommended amounts (>10 standard glasses per week or > 2 standard glasses per day).
20. Subject living in the same home as a subject currently participating in this evaluation.
21. Subjects defined as individuals whose willingness to volunteer in the clinical trial may be unduly influenced by benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. (Examples are members of a group with a hierarchical structure linked to the Investigator or to the Sponsor, such as students, subordinate hospital and laboratory personnel, employees of the Investigator or of the Sponsor, relatives of the Sponsor).
22. Employees and/or children/family members or relatives of employees of Danone Global Research & Innovation Center or the participating sites.
23. Belonging to a population covered by articles L.1121-6 (persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care), and L.1121.8 (adults under legal protection or unable to express their consent) of the CSP (French Public Health Code).
24. Subjects admitted to a health or social care facility.
25. Individuals with a known case of diabetes mellitus (type 1 or type 2), or those with a known HbA1c ≥ 6.5% at screening, or currently receiving antidiabetic treatment (oral or injectable).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Non-tolerance | After 7 days of study product consumption
  Percentage of non-tolerance events as defined by participant dropping out due to digestive symptoms during the 7-day intervention phase
Score of the Digestive Symptoms Frequency Questionnaire (DSFQ) | After 7 days of study product consumption
  The absolute change from baseline to day 7 of the intervention phase on the total score of the Digestive Symptoms Frequency Questionnaire (DSFQ)

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) score | After 7 days of study product consumption
  The absolute change of digestive symptoms from baseline to day 7 of the intervention phase on the daily Visual Analog Scale (VAS) score
Maximum score of digestive symptoms | After 7 days of study product consumption
  The maximum score of digestive symptoms from baseline to day 7 of the intervention phase using the daily Visual Analog Scale (VAS)
The time to maximum score of digestive symptoms | After 7 days of study product consumption
  The time to maximum score of digestive symptoms (Tmax) on the daily Visual Analog Scale (VAS) from baseline to day 7 of the intervention phase
incremental Area Under Curve (iAUC) | After 7 days of study product consumption
  The daily Visual Analog Scale (VAS) score incremental Area Under Curve (iAUC) from baseline to day 7 of the intervention phase
Digestive Symptoms Frequency Questionnaire (DSFQ) | After 7 days of study product consumption
  The absolute change from baseline to day 7 of the intervention phase on individual symptoms scores (4 symptoms sub-scores) of the Digestive Symptoms Frequency Questionnaire (DSFQ)
Daily VAS at run-in phase | After 7 days without product consumption
Stool Frequency Questionnaires (SFQ) at run-in phase | After 7 days without product consumption
Bristol Stool Scale (BSS) at run-in phase | After 7 days without product consumption
Food Frequency Questionnaire (FFQ) at V3 | After 7 days without product consumption
Nutrient daily intake and food group daily intake (MyFood24) at run-in phase | After 7 days without product consumption
FODMAP daily content (Monash calculator) at run-in phase | After 7 days without product consumption
DSFQ (total score and the 4 symptom sub-scores) at the run-in phase | After 7 days without product consumption
Rome IV at V1 (IBS, FB, U-FBD, abdominal pain, bloating/distention at least once a week) | At inclusion
Breath hydrogen concentration (ppm - OMED health device by Owlstone Medi-cal) from baseline (run-in) to day 7 of the intervention phase | After 7 days of study product consumption
Breath methane concentration (ppm - OMED health device by Owlstone Medi-cal) from baseline (run-in) to day 7 of the intervention phase | After 7 days of study product consumption
Association between breath hydrogen and methane concentrations and DSFQ score | After 7 days of study product consumption
Association between breath hydrogen and methane concentrations and VAS score | After 7 days of study product consumption

CONTACTS AND LOCATIONS:
Locations (1):
- CEN experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: No